CLINICAL TRIAL: NCT03535233
Title: Combined Topical 5% Minoxidil and Potent Topical Corticosteroid Versus Intralesional Corticosteroid in the Treatment of Alopecia Areata A Randomized Controlled Trial
Brief Title: Topical 5% Minoxidil and Potent Topical Corticosteroid Versus Intralesional Corticosteroid in the Treatment of Alopecia Areata
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona El-Kalioby, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AA22
Record Dates: First submitted 2018-05-11; First posted 2018-05-24 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Alopecia Areata
Keywords: Alopecia areata, intralesional corticosteroid, minoxidil, clobetasol propionate, IL-23, TGFβ-1
MeSH Terms: conditions — Alopecia Areata | interventions — Triamcinolone Acetonide; Minoxidil; Clobetasol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intralesional group (Active Comparator): intralesional triamcinolone acetonide 5 mg/ml monthly
  Interventions: Drug: Triamcinolone Acetonide
- Topical therapy group (Active Comparator): Minoxidil 5% topical solution applied twice daily and topical clobetasol propionate 0.05% cream applied once daily every night
  Interventions: Drug: Minoxidil 5 % Topical Spray; Drug: clobetasol propionate

INTERVENTIONS:
Drug: Triamcinolone Acetonide
  Arms: Intralesional group
Drug: Minoxidil 5 % Topical Spray
  Arms: Topical therapy group
Drug: clobetasol propionate
  Arms: Topical therapy group

SUMMARY:
Alopecia areata (AA) presents with circumscribed patches of non-scarring hair loss. It inflects a significant psychological and social burden. Many treatment options are used for the treatment of AA. Randomized controlled trials comparing intralesional and topical therapy and comparing combinations are few.

The aim of this work is to evaluate the efficacy of combined topical 5% minoxidil and potent topical corticosteroid therapy compared to intralesional triamcinolone injection in alopecia areata

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with scalp alopecia areata, patchy type, of at least 2 months duration.

Exclusion Criteria:

* Alopecia totalis and alopecia universalis.
* Alopecia areata solely affecting the beard.
* Pregnant and lactating.
* Patients known to have autoimmune diseases e.g. autoimmune thyroid disease, vitiligo or SLE.
* Patients receiving systemic treatment relevant to alopecia areata within 3 months before enrollment into the study or topical treatment relevant to alopecia areata within 2 months before.
* Patients with a dermatological condition affecting the scalp other than AA: e.g. psoriasis, eczema.
* Patients with psychiatric illness or psychological state interfering with compliance or influencing the expectation of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Clinical assessment using SALT score (Severity of Alopecia Tool score) | 3 months
  SALT score is a quantitative assessment scale for the evaluation of percentage of scalp hair loss.
  The percent surface area of each of the 4 scalp is determined: Vertex (top): 40% (0.4) of scalp surface area; each side of scalp (right and left profile): each 18% (0.18) of scalp surface area; posterior aspect (back) of scalp: 24% (0.24) of scalp surface area. The percentage of hair loss in any of these 4 aspects is calculated as the percentage of hair loss multiplied by percent surface area of the scalp in that area. SALT score is the sum of product of each section in the above mentioned areas. SALT score is calculated before and after therapy.
  Lowest value: 0%: indicates abscence of clinical disease, Highest value: 100%: indicate 100% affection of the scalp

SECONDARY OUTCOMES:
Dermoscopic evaluation | 3 months
  Dermoscopic assessment of the scalp is performed using DermaLite II Pro HR dermoscope, Germany.
  Dermoscopic examination is graded according to a scale provided by Trink and colleagues (2013).
  The percentage of dystrophic hairs was evaluated on a 4-point scale as followed:
  * 3= >50% dystrophic hairs
  * 2 = 30-50% dystrophic hairs
  * 1 = 1-29% dystrophic hairs
  * 0 = no dystrophic hairs
Quantitative measurement of Transforming growth factor-beta 1 (TGF-β1) | 3 months
  ELISA
Quantitative measurement of Interleukin-23 (IL-23) | 3 months
  ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Nermine H El-Eishi, MD, Study Chair — Cairo University; Heba M Mashaly, MD, Principal Investigator — Cairo University; Solwan I El-Samanoudy, MD, Principal Investigator — Cairo University; Mona MI ElKalioby, MD, Principal Investigator — Cairo University; Olfat G Shaker, MD, Principal Investigator — Cairo University; Rania M Abdel-Hay, MD, Principal Investigator — Cairo University